CLINICAL TRIAL: NCT02630914
Title: Medical and Surgical Hybrid Treatment of Atrial Fibrillation: Epicardial and Endocardial Combined Approach.
Brief Title: Medical and Surgical Hybrid Treatment of Atrial Fibrillation.
Acronym: HT2AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/14/7424
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2018-12

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Epicardial surgical removal; Closure of the left atrial; Left atrial appendage (LAA)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): All patients will have the hybrid procedure of ablation of atrial fibrillation.
  Interventions: Device: The AtriCure Synergy Ablation System

INTERVENTIONS:
Device: The AtriCure Synergy Ablation System — The AtriCure Synergy Ablation System will be used on all patients for AF ablation.

SUMMARY:
The objective of the study is to investigate the feasibility of a hybrid procedure removal of the atrial fibrillation.

This is a single procedure for both surgical epicardial by minimally invasive route (Thoracoscopy) without even flow controlled and supplemented if necessary by extra corporeal intracavitary route at the same time.

This faster procedure combined with complete lesions have a higher success rate and less frequent re-hospitalizations of patients.

ELIGIBILITY:
Inclusion Criteria:

patients with complex AF defined by the following criteria :

* AF> 1 week or long term persistent> 1 year
* AND Symptomatic
* AND after failure of treatment of anti-arrhythmic or against-indication for anti-arrhythmic

Exclusion Criteria:

The exclusion criteria are relevant contraindications thoracoscopy or the non-complex nature of the AF:

* Paroxysmal AF or AF cardioverted anti-arrhythmic test (unless against indicated)
* Recent AF for which a simple gesture is intracavitary considered sufficient
* Permanent AF
* Asymptomatic AF
* Very old AF (> 5 years) or atrial major ectasia (> 60 mm)
* Need another surgery (valve bypass coronary)
* Previous history of sternotomy or thoracotomy
* High-risk surgical or anesthetic Patient
* BMI> 35
* Sleep Apnea
* Ejection fraction <35%
* Thoracic trauma history
* Veins Pulmonary stenosis> 50%
* Hyperthyroidism
* Thrombus in LAA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with complete procedure or not | 3 hours
  At the end of the intervention, the doctor evaluates whether the procedure was complete with electric exclusion of the posterior wall of the left atrium and the 4 pulmonary veins.

SECONDARY OUTCOMES:
Number of atrial fibrillation episode | 12 months
Stroke Rate | 12 months
Hospitalization for heart failure | 12 months
  The number of hospitalizations for heart failure after hybrid procedure
Evaluation of Quality of life (EQ-5D according to the survey-3L) | 12 months
  The quality of life will be measured using the EQ-5D 3L questionnaire (EQ-5D according to the survey-3L)
The cost-effectiveness ration | 12 months
  Cost estimates will be conducted from the perspective of health insurance. The expenses incurred in the care of patients will be counted during the follow-up year.
  The effectiveness will be assessed against the complications of strategy

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Marcheix, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, Midi Pyrenees, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rollin A, Mandel F, Grunenwald E, Mondoly P, Monteil B, Marcheix B, Maury P. Hybrid surgical ablation for persistent or long standing persistent atrial fibrillation: A French single centre experience. Ann Cardiol Angeiol (Paris). 2020 Apr;69(2):86-92. doi: 10.1016/j.ancard.2020.03.008. Epub 2020 Mar 30. PMID 32241522